CLINICAL TRIAL: NCT01117233
Title: A Randomised, Placebo Controlled, Double-Blind, Third Party Open, Parallel Group Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-04427429 Administered Intravenously To Healthy Adult Volunteers
Brief Title: Study In Healthy Adult Volunteers To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-04427429
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B0141002
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Healthy volunteers; PK; PD; safety and toleration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Single IV Dose 1 (Experimental)
  Interventions: Drug: PF-04427429
- Single IV Dose 2 (Experimental)
  Interventions: Drug: PF-04427429
- Single IV Dose 3 (Experimental)
  Interventions: Drug: PF-04427429
- Single IV Dose 4 (Experimental)
  Interventions: Drug: PF-04427429
- Single IV Dose 5 (Experimental)
  Interventions: Drug: PF-04427429

INTERVENTIONS:
Drug: PF-04427429 — single intravenous infusion of 10 mg PF-04427429 or placebo
  Arms: Single IV Dose 1
Drug: PF-04427429 — single intravenous infusion of 30 mg PF-04427429 or placebo
  Arms: Single IV Dose 2
Drug: PF-04427429 — single intravenous infusion of 100 mg PF-04427429 or placebo
  Arms: Single IV Dose 3
Drug: PF-04427429 — single intravenous infusion of 300 mg PF-04427429 or placebo
  Arms: Single IV Dose 4
Drug: PF-04427429 — single intravenous infusion of 1000 mg PF-04427429 or placebo
  Arms: Single IV Dose 5

SUMMARY:
The purpose is to study the safety, tolerability, pharmacokinetics and pharmacodynamics of PF-04427429 administered intravenously to healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 50 years inclusive (unless local regulations dictate a minimum age of 21 years). Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight of between 50 kg and 100 kg inclusive.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, genitourinary, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, symptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption.
* 12-lead ECG demonstrating QTcF >450 msec at Screening. If QTcF exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTcF values should be used to determine the subject's eligibility.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Adverse events, Vitals, ECG, laboratory safety tests, IV infusion site reaction | up to 84 days
Plasma pharmacokinetics of PF-04427429 | up to 84 days

SECONDARY OUTCOMES:
Free and total CGRP plasma concentrations | up to 84 days
anti-drug antibody | up to 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0141002&StudyName=Study%20In%20Healthy%20Adult%20Volunteers%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20PF-04427429